CLINICAL TRIAL: NCT05501639
Title: Exacerbation Risk in Asthma
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 0205-0547
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Results first posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2023-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- tiotropium + inhaled corticosteroids (ICS) group
  Interventions: Drug: tiotropium; Drug: inhaled corticosteroids (ICS)
- long-acting β2-agonists (LABA) + inhaled corticosteroids (ICS) group
  Interventions: Drug: long-acting β2-agonists (LABA); Drug: inhaled corticosteroids (ICS)

INTERVENTIONS:
Drug: tiotropium — tiotropium
  Groups: tiotropium + inhaled corticosteroids (ICS) group
Drug: long-acting β2-agonists (LABA) — long-acting β2-agonists (LABA)
  Groups: long-acting β2-agonists (LABA) + inhaled corticosteroids (ICS) group
Drug: inhaled corticosteroids (ICS) — inhaled corticosteroids (ICS)

SUMMARY:
The purpose of this study is to conduct a comparative analysis of patients using Tiotropium in combination with Inhaled Corticosteroids (ICS) versus those that use long-acting β2-agonists (LABA) medication in combination with ICS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with least two asthma diagnosis
* Patients will be required to be concurrently on inhaled corticosteroids (ICS)+Tiotropium (tio) (specifically Tiotropium Respimat® 1.25 mcg) or ICS/LABA
* Patients will be required to have enrollment for at least 6 months prior to ICS+Tio or ICS/LABA use

Exclusion Criteria:

* Patients with least two diagnosis of chronic obstructive pulmonary disease (COPD) at any time during the study period
* Patients less than 12 years of age
* Patients on biologics within 6 months prior to ICS+Tio or ICS/LABA use
* Patients with prior Tio or ICS/LABA use during the 6-month baseline period
* Patients with urinary bladder obstruction, urinary retention, and glaucoma
* After the propensity score matching (PSM) process, unmatched patients

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with least two asthma diagnosis will be included. Patients will be required to have enrollment for at least 6 months prior to ICS+Tio or ICS/LABA use.
Sampling Method: Non-Probability Sample
Enrollment: 1899 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- eMax Health, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The objective of this study was to conduct a retrospective cohort study comparing asthma patients taking tiotropium in combination with inhaled corticosteroids (ICS) versus patients taking long-acting β2-agonists (LABA) medication in combination with ICS.
Pre-assignment Details: Propensity score matched (PSM) cohorts of patients between the ICS + tiotropium (tio) and ICS/LABA groups. Patients >=12 years with least two asthma diagnosis were included and be required to be concurrently on ICS + tio or ICS/LABA.
Groups:
- Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort: Patients with at least two asthma diagnosis who were treated concurrently with inhaled corticosteroids (ICS) + tiotropium (specifically tiotropium Respimat 1.25 mcg) between 2014 and 2020. Patients were matched to patients receiving inhaled corticosteroids (ICS) + long-acting β2-agonists (LABA) using a time-conditional propensity score-matched approach.
- Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort: Patients with at least two asthma diagnosis who were treated concurrently with inhaled corticosteroids (ICS) + long-acting β2-agonists (LABA) between 2014 and 2020. Patients were matched to patients receiving inhaled corticosteroids (ICS) + tiotropium (specifically tiotropium Respimat 1.25 mcg) using a time-conditional propensity score-matched approach.
Period: Overall Study
Arm/Group | Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort | Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort
Started | 633 | 1266
Completed | 633 | 1266
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The main analysis was on matched cohorts of patients between the ICS + tio and ICS/LABA cohorts using a 1:2 propensity score matching (PSM) approach. PSM resulted in a match of each ICS + tio patient to 2 ICS/LABA patients. Baseline measures were presented for matched populations.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort | Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort | Total
Number analyzed (Participants) | 633 | 1266 | 1899
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.00 (16.43) | 46.14 (16.30) | 45.94 (16.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 453 | 903 | 1356
  Male | 180 | 363 | 543
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Race and Ethnicity were not collected from any participant. Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time to First Severe Exacerbation
Description: Severe exacerbation defined as:
  * Hospitalization with primary diagnosis of asthma or
  * Emergency room (ER) visit with primary diagnosis of asthma The analysis of this endpoint is based on number of observations (exacerbations).
  Index date is defined as date when patient entered the cohort. Design 1: A time-varying covariate approach to classify drug exposure time for each comparator drug during follow up was used. For each individual study drug, medication exposure + non-exposure windows during the follow-up time for each medication were identified/defined using date of prescription filled + days' supply listed on prescription claim + 50% additional days.
Time Frame: From index date to first severe exacerbation, up to 1 year.
Population: The main analysis was on matched cohorts of patients between the ICS + tio and ICS/LABA cohorts using a 1:2 propensity score matching (PSM) approach. PSM resulted in a match of each ICS + tio patient to 2 ICS/LABA patients. Values were presented for matched populations. Only patients with severe exacerbation were included in this analysis.
Measure: Mean (Standard Deviation); unit: Days
Units Other Than Participants: observations
Arm/Group | Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort | Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort
Number analyzed (Participants) | 4 | 23
Number analyzed (observations) | 4 | 23
Days | 43.75 (30.50) | 49.43 (34.07)
Statistical Analysis 1: Comparison: Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort vs Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort; Test type: Other; p = 0.758, Log Rank

2. Secondary Outcome: Time to First Moderate-or-severe Exacerbation
Description: as for outcome 1
Time Frame: From index date to first moderate-or-severe exacerbation, up to 1 year.
Population: The main analysis was on matched cohorts of patients between the ICS + tio and ICS/LABA cohorts using a 1:2 propensity score matching (PSM) approach. PSM resulted in a match of each ICS + tio patient to 2 ICS/LABA patients. Values were presented for matched populations. Only patients with moderate-to-severe exacerbation were included in this analysis.
Measure: Mean (Standard Deviation); unit: Days
Units Other Than Participants: observations
Arm/Group | Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort | Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort
Number analyzed (Participants) | 99 | 335
Number analyzed (observations) | 99 | 335
Days | 65.8 (85.88) | 58.88 (83.98)
Statistical Analysis 1: Comparison: Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort vs Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort; Test type: Other; p = 0.474, Log Rank

3. Secondary Outcome: Percentage of Patients With Exacerbation
Description: Percentage of patients with exacerbation is presented. Design 2: The second analysis, included on an ad-hoc basis was using an intent-to-treat (ITT) design where patients were assigned to the cohort, they were part of at the index date.
Time Frame: From index date through first report of exacerbation, up to 1 year.
Population: The main analysis was on matched cohorts of patients between the ICS + tio and ICS/LABA cohorts using a 1:2 propensity score matching (PSM) approach. PSM resulted in a match of each ICS + tio patient to 2 ICS/LABA patients. Values were presented for matched populations.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort | Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort
Number analyzed (Participants) | 633 | 1266
Percentage of Participants
  Severe exacerbation | 3.8 | 3.2
  Moderate-or-severe exacerbation | 50.1 | 45.3
Statistical Analysis 1: Comparison: Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort vs Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort; Test type: Other; p = 0.472, Chi-squared

4. Secondary Outcome: Rate of Exacerbation at 6 Months and One Year
Description: Rate of exacerbation at 6 months and one year is presented.
Time Frame: at 6 months and one year
Population: as for outcome 3
Measure: Number; unit: Events per 100 person years
Arm/Group | Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort | Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort
Number analyzed (Participants) | 633 | 1266
Events per 100 person years
  At 6 months | 3.21 | 4.96
  At one year | 4.46 | 4.45
Statistical Analysis 1: Comparison: Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort vs Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort; Test type: Other; Incidence rate ratio = 0.647, 95% CI 2-sided [0.261 to 1.604] — Incidence rate ratio at 6 months
Statistical Analysis 2: Comparison: Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort vs Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort; Test type: Other; Incidence rate ratio = 1.005, 95% CI 2-sided [0.513 to 1.969] — Incidence rate ratio at 12 months

5. Secondary Outcome: Percentage of Patients With Health Care Resource Utilization (HCRU)
Description: Percentage of patients with Health care resource utilization (HCRU) is presented and is defined as hospitalizations, emergency room (ER) visits, and outpatient visits during follow-up, all-cause and asthma related.
Time Frame: From index date to end of follow-up, up to 1 year.
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort | Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort
Number analyzed (Participants) | 633 | 1266
Percentage of Participants
  Hospitalisations | 7 | 9
  Asthma-related hospitalisations | 1 | 1
  Emergency department (ED) visits | 23 | 21
  Asthma-related ED visits | 3 | 2
  outpatient (OP) visits | 96 | 95
  Asthma-related OP visits | 64 | 54
Statistical Analysis 1: Comparison: Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort vs Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort; Hospitalisations; Test type: Other; p = 0.222, Chi-squared
Statistical Analysis 2: Comparison: Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort vs Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort; Asthma-related hospitalisations; Test type: Other; p = 0.553, Chi-squared
Statistical Analysis 3: Comparison: Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort vs Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort; ED visits; Test type: Other; p = 0.192, Chi-squared
Statistical Analysis 4: Comparison: Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort vs Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort; Asthma-related ED visits; Test type: Other; p = 0.383, Chi-squared
Statistical Analysis 5: Comparison: Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort vs Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort; OP visits; Test type: Other; p = 0.338, Chi-squared
Statistical Analysis 6: Comparison: Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort vs Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort; Asthma-related OP visits; Test type: Other; p < 0.0001, Chi-squared

6. Secondary Outcome: Health Care Resource Utilization (HCRU)
Description: Health care resource utilization (HCRU) are presented including frequency of hospitalizations, ER visits, outpatient visits. Outpatient visits are defined as clinic, hospital, or other medical institution (e.g. public health, etc.) visit as an outpatient.
  Mean and standard deviations of:
  * Number of hospitalisations per person per month
  * Number of asthma-related hospitalisations per person per month
  * Number of ER visits per person per month
  * Number of asthma-related ER visits per person per month
  * Number of outpatient visits per person per month
  * Number of asthma-related outpatient visits per person per month are presented.
Time Frame: From index date to end of follow-up, up to 1 year.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Count of HCRU per person per month
Arm/Group | Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort | Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort
Number analyzed (Participants) | 633 | 1266
Count of HCRU per person per month
  Hospitalisations | 0.007 (0.051) | 0.009 (0.049)
  Asthma-related hospitalisations | 0.001 (0.015) | 0.001 (0.017)
  Emergency department (ED) visits | 0.035 (0.131) | 0.032 (0.139)
  Asthma-related ED visits | 0.002 (0.019) | 0.002 (0.018)
  Outpatient (OP) visits | 1.804 (1.836) | 1.343 (1.462)
  Asthma-related OP visits | 0.130 (0.218) | 0.096 (0.226)
Statistical Analysis 1: Comparison: Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort vs Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort; Hospitalisations; Test type: Other; p = 0.538, t-test, 2 sided
Statistical Analysis 2: Comparison: Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort vs Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort; Asthma-related hospitalisations; Test type: Other; p = 0.913, t-test, 2 sided
Statistical Analysis 3: Comparison: Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort vs Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort; ED visits; Test type: Other; p = 0.688, t-test, 2 sided
Statistical Analysis 4: Comparison: Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort vs Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort; Asthma-related ED visits; Test type: Other; p = 0.892, t-test, 2 sided
Statistical Analysis 5: Comparison: Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort vs Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort; OP visits; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 6: Comparison: Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort vs Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort; Asthma-related OP visits; Test type: Other; p = 0.002, t-test, 2 sided

7. Secondary Outcome: Percentage of Patients With Use of Rescue Medications
Description: Percentage of patients with use of rescue medications is presented. Use of rescue medication is defined as patients with one or more short-acting β2-agonists (SABA) claims during the follow-up period.
Time Frame: From index date to end of follow-up, up to 1 year.
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort | Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort
Number analyzed (Participants) | 633 | 1266
Percentage of Participants | 57 | 55
Statistical Analysis 1: Comparison: Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort vs Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort; Test type: Other; p = 0.378, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse event information was not applicable for this study.
Description: This was an observational study and was not designed to assess adverse event; therefore safety reporting was not applicable for this study. Adverse events were not planned to be collected as defined in the study protocol. Adverse Events were not monitored/assessed.
Arm/Group | Tiotropium (Tio) + Inhaled Corticosteroids (ICS) Cohort | Long-acting β2-agonists (LABA) + Inhaled Corticosteroids (ICS) Cohort
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT05501639/Prot_SAP_000.pdf